CLINICAL TRIAL: NCT07164508
Title: Revolutionizing Adapted Physical Activity for Individuals With Physical Disabilities: Examining the Health Impact of and Promoting Sitting Light Volleyball in the Greater Bay Area
Brief Title: Examining the Health Impact of and Promoting Sitting Light Volleyball in the Greater Bay Area
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: The Hong Kong Society for Rehabilitation (Other)
Responsible Party: Principal Investigator, LEUNG Ka Man Carman, Associate Professor, Principal Investigator, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R8003-25
Record Dates: First submitted 2025-08-15; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Physial Disabilities
Keywords: Physical Impairments; Adapted Sports; Adults; Hong Kong; Mainland China

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Independent evaluators assessing participants' outcomes, and those involved in data entry and analysis will be blinded to group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sitting Light Volleyball Intervention Group (Active Comparator): 75 randomly selected participants within the demographic of adults with physical disabilities who will undergo a 16-week Sitting Light Volleyball intervention, comprised of 32 training sessions with 2 x 75-minute sessions per week, according to the World Health Organization recommendations. This intervention plan is based on the research team's previous Sitting Light Volleyball program designed for people with physical disabilities, and will cover basic Sitting Light Volleyball skills and posture, team tactics, as well as rules and regulations.
  Interventions: Behavioral: Sitting Light Volleyball Intervention
- Group Seated Dance Intervention Group (Active Comparator): 75 randomly selected participants within the demographic of adults with physical disabilities who will undergo a 16-week group Seated Dance intervention, comprised of 32 training sessions with 2 x 75-minute sessions per week, according to the World Health Organization recommendations. Participants in this group will learn freestyle para-dance in a group setting, including hip-hop and Latin dance. They will practice step sequences of increasing complexity whilst seated, and later, music will be added to their dance routines.
  Interventions: Behavioral: Group Seated Dance Intervention
- Control Group (No Intervention): 75 randomly assigned participants in this group will be instructed to maintain their normal daily activities, and will be asked to join monthly non-exercise social gatherings (e.g. health talks) to balance the psychosocial effects associated with the regular gatherings in the other groups.

INTERVENTIONS:
Behavioral: Sitting Light Volleyball Intervention — 16-week intervention centered around Sitting Light Volleyball, an adaptive sport developed by the Project Coordinator specifically for adults with physical disabilities.
  Arms: Sitting Light Volleyball Intervention Group
Behavioral: Group Seated Dance Intervention — 16-week intervention program for adults with physical disabilities centered around para dance in a group setting of various dance styles.
  Arms: Group Seated Dance Intervention Group

SUMMARY:
The present study builds on the promising result of our SLVB pilot study with the aim to extend the works' impact by investigating the effectiveness of a SLVB intervention on the physical and psychological health outcomes in adults with physical disabilities in HKG by collecting quantitative and qualitative data in a larger sample (225 participants). The investigators hypothesize that the SLVB and Seated Dance (SD) interventions will improve physical and psychological health outcomes, and quality of life compared to the control group, with SLVB expected to be more effective than SD in enhancing health outcomes for PWPDs. Using the consolidated evidence on the benefits of SVLB from our research work, the investigators will promote SLVB in HKD and CHN by organizing i) train-the-trainer workshops (325 trainers trained), ii) SLVB classes (about 1270 PWPD in HKG and CHN) and iii) SLVB competitions in HKG and CHN (initial rounds of competition will be held across Hong Kong, Shenzhen and Guangzhou, with the finals to be held in Hong Kong, totaling to 408 participants). The investigators combine the evidenced benefits of SVLB with the Train-The-Trainer approach, suggested by the World Health Organization, to achieve community engagement and it is regarded as a solution to institutional barriers in promoting adapted physical activity. SLVB teaching aids will also be developed to promote the activities.

DETAILED DESCRIPTION:
One hundred and thirty-eight participants will be randomly assigned into the SLVB, Seated Dance (SD), and control groups in a 1:1:1 ratio. Outcome assessors will be blinded to treatment allocation. Data will be collected at baseline (pretest), after a 16-week intervention (posttest), at 3 months and 6 months after the intervention. Both the SLVB and SD intervention programmes consist of 32 training sessions, with 2 x 75- min sessions per week. The duration of the proposed intervention is consistent with the recommendation of World health Organization. The SLVB intervention programme will be based on our previous SLVB programme specifically designed for PWPD. Programme content will include SLVB basic skills and posture, basic team tactics, and rules and regulations. In the SD group, participants will learn freestyle para dance in sessions, including hip-hop and Latin dance. They will learn step sequences of increasing complexity in a seated position, and music will then be added. Participants in the control group will be instructed to maintain their normal daily activity and asked to join monthly non-exercise social gatherings (e.g., health talk) to balance the psychosocial effect of the regular gatherings in other groups. Inclusive criteria for participants will be (a) aged ≥18 years; (b) PWD registered in the Central Registry for Rehabilitation; (c) diagnosed with physical disabilities such as impaired muscle power, limb deficiency, or leg length difference, using the SVB and Para dance classification of International Paralympic Committee; (d) with at least one functional arm; (e) with a normal to mild grade intellectual disability; (f) have not participated in a structured PA programme during the 6 months preceding the study; and (g) can communicate in Chinese. The Mini-Mental Statewill be used to screen for abnormal cognitive function; the Berg Balance Scale will be used to screen for participant's sitting balance ability. Participants who a) record an MMSE score ≤ 17; b) are unable to sit unsupported [balance score ≤ 2 (i.e., sit 30 seconds)]; c) Body Mass index (BMI) ≥ 27; d) have had orthopaedic surgery 6 months prior to the study entry; e) have a history of cardiovascular disease that hinders study participation; f) have seeing and/or hearing difficulties; g) have not been approved by his/her physician to participate in the study due to a limiting medical condition, will be excluded from the study. Based on a more conservation effect size (Cohen's d = .6) from the physical attributes of our previous SLVB intervention study, a total sample of 111 PWPD (with 20% expected dropout rate) is required in this study to achieve power of 80% at p ≤ .05. The investigators, therefore, aim to recruit a total sample size of 138 participants (46 participants per NGO serving PWPD, 3 NGOs are needed) and allocated in a 1:1:1 ratio into SLVB, SD and control groups (15-16 participants in each arm in each NGO). Procedures. Participants will be recruited through recruitment talk(s) conducted by the research team and by advertisements in the partnered NGOs. First, an initial information session will be delivered to groups of potential participants by providing them with intervention details and distributing the informed consent statement. After obtaining the participant's signed informed consent, data collection will be conducted by the SRA and trained student helpers. Before the pretest, participants will undergo screening tests such as MMSE. In addition to completing questionnaires, participants will begin by taking fitness and other tests according to the standardized testing protocol. Next, an independent researcher, not otherwise involved in the study, will use a computer-based random number generator to randomly assign participants into SLVB, SD, or control groups. The intervention will begin next week. Participants will complete a posttest and follow-up tests upon completion of the 16-week intervention, 3 and 6 months after the intervention, respectively, using procedures identical to those described for the pretest measurements. The independent evaluators assessing the participants' outcomes and individuals performing data entry and data analysis will be blinded to group assignment.

Measures (Primary - Physical health outcomes) i. Physical fitness. The Brockport physical fitness test will be used to measure the physical fitness of participants. The fitness tests include a grip test (upper body muscular strength), dumbbell press test (upper body muscular endurance), skinfold test and body mass index evaluation (body composition), and shoulder stretch test (flexibility). Submaximal arm ergometry test, six-Minute Arm Test will be used to measure participant's aerobic endurance. The validity and reliability of the above tests have been confirmed for use with PWD and it has been used in HK.

ii. Sitting balance. A modified Functional Reach Test will be used to assess limits of stability by measuring the maximum distance that an individual can reach forward and laterally while sitting in a fixed position. Its reliability and validity have been supported for adults with disabilities.

iii. Anticipation time. A Bassin Anticipation Timer (BAT, Lafayette Instrument Company, Model 35575) will measure the participant's visual acuity related to eye-hand coordination and anticipation (in milliseconds.). Using BAT devices, participants will be instructed to press a button to coincide with light arrival at the target.

Measures (Secondary - Psychological health outcomes) i. Quality of life (QoL). QoL will be measured using a shortened version of the SF36 Health Survey (SF-12). Reliability and validity have been evaluated in Chinese. SF-12 comprises eight domains such as mental health, social, and physical functioning …etc.

ii. PA enjoyment. A short version of the Physical Activity Enjoyment Scale (PACES) in Chinese will be used to measure PA enjoyment in the study. Other studies have also validated the psychometric properties of this 8-item PACES.

ii. Mindful self-care. Mindful Self-Care Scale - Chinese Version (24 item) measures an individual's level of mindful self-care across various dimensions, including physical care, supportive relationships, mindful awareness, self-compassion and purpose, mindful relaxation, and supportive structure.

Data analysis. Intent-to-treat sample will be used in the primary analysis. The Generalized Estimating Equation (GEE) model will be used to test the statistical significance of the mean changes in the primary and secondary outcomes among the three groups. Adjustments will be performed for the age and gender of the participants. The GEE model handles the auto-correlations among the repeated measurements within a participant in each group, as well as non-normal data, and accommodates missing data points across the measurement time points. The same statistical analysis will be performed in the per-protocol sample as a secondary analysis. A dose-response analysis will be conducted by treating adherence to the intervention as an independent variable. Data will be analyzed using SPSS 27.0 with a significance level set at .05 Qualitative study is used to determine the barriers and facilitators of the intervention implementation from the perspective of stakeholders, thirty participants in the SLVB group will be recruited using purposive sampling, stratified by gender and completion of our intervention. Intervention completion is defined as an attendance rate of 80% or higher. Next, 6 administrators and 6 coaches will also be invited to participate in the interview. This sample size is referenced to a similar study using the Consolidated Framework for Implementation Research (CFIR) in PWD, qualitative research meta-synthesis in PWPD's PA and our previous SLVB qualitative studies. Procedures. Participants (group of five for participants, group of two for administrators, group of two for coaches) in the SLVB group will be invited to join this qualitative arm. It is guided by our SLVB qualitative studies and the CRIF, which provides 39 constructs housed in 5 domains such as intervention characteristics, and implementation process. CFIR will guide this study's data collection, analysis and reporting.

In terms of data analysis, all interviews will be transcribed verbatim and coded using QSR-NVivo. Using thematic analysis, data will be organized into themes based on CFIR. Two independent coders will read, re-read, and code the interview transcripts to ensure that coding is done following the CFIR coding guide. Finally, coded transcripts will be compared, followed by another discussion with the coders and investigators to facilitate further the development of themes related to the framework. The 32-point consolidated criteria for reporting qualitative studies will be used to report the result.

ELIGIBILITY:
Inclusion Criteria:

* People with disabilities registered in the Central Registry for Rehabilitation.
* Diagnosed with physical disabilities such as impaired muscle power, limb deficiency, or leg length difference, using the soft volleyball and Para dance classification of International Paralympic Committee.
* Has at least one functional arm.
* With a normal to mild grade intellectual disability.
* Have not participated in a structured physical activity program during the 6 months preceding the study.
* Can communicate in Chinese.

Exclusion Criteria:

* Having a recorded Mini-Mental State Examination score of 17 or below.
* Unable to sit unsupported, by recording a balance score at or below 2 on the Berg Balance Scale (indicating they are able to sit for a maximum of 30 seconds).
* Having a Body Mass Index of 27 or above.
* Have had orthopedic surgery 6 months (or less) prior to the study entry.
* Have a history of cardiovascular disease that hinders study participation.
* Have seeing and/or hearing difficulties.
* Have not been approved by his/her physician to participate in the study due to a limiting medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical fitness - Physical health outcome - Muscular Strength | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  The Brockport Physical Fitness Test will be used to assess multiple components of physical fitness in participants. This includes Upper Body Muscular Strength: Assessed using the Grip Test, reported in kilograms.
Physical fitness - Physical health outcome - Muscular Endurance | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  The Brockport Physical Fitness Test will be used to assess multiple components of physical fitness in participants. This includes Upper Body Muscular Endurance. it will be assessed using the Dumbbell Press Test, reported as number of repetitions.
Physical fitness - Physical health outcome - Body Composition - Body Mass Index | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  The Brockport Physical Fitness Test will be used to assess multiple components of physical fitness in participants. This includes Body Composition. Body Mass Index. Weight and height will be combined to report BMI in kg/m^2.
Physical fitness - Physical health outcome -The Brockport Physical Fitness Test | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  The Brockport Physical Fitness Test will be assessed using the Skinfold Test (reported in millimeters)
Physical fitness - Physical health outcome - Flexibility | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  The Brockport Physical Fitness Test will be used to assess multiple components of physical fitness in participants. This includes flexibility, assessing using the Shoulder Stretch Test, reported as pass/fail based on reach criteria.
Physical fitness - Physical health outcome - Aerobic Endurance | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  The Brockport Physical Fitness Test will be used to assess multiple components of physical fitness in participants. This includes Aerobic Endurance. It will be assessed using the Submaximal Arm Ergometry Test and the Six-Minute Arm
Anticipation time - Physical health outcome | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  A Bassin Anticipation Timer (BAT, Lafayette Instrument Company, Model 35575) will measure the participant's visual acuity related to eye-hand coordination and anticipation (in milliseconds.). Using BAT devices, participants will be instructed to press a button to coincide with light arrival at the target.
Sitting balance - Physical health outcome | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  A modified Functional Reach Test will be used to assess limits of stability by measuring the maximum distance that an individual can reach forward and laterally while sitting in a fixed position. Its reliability and validity have been supported for adults with disabilities.

SECONDARY OUTCOMES:
Quality of life - Psychological health outcome | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  Quality of life will be measured using a shortened version of the Short Form (12) Health Survey. Reliability and validity have been evaluated in Chinese. The survey comprises eight domains such as mental health, social, and physical functioning …etc. It will be scored in a 5-point Likert scale (1=often, 5=never), with some reversely asked questions. After reverse-scoring the negatively worded items, a higher total score means better life quality.
Physical Activity Enjoyment - Psychological health outcome | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  A short version of the Physical Activity Enjoyment Scale in Chinese will be used to measure physical activity enjoyment in the study. Chung and the primary investigator of this study have also validated the psychometric properties of this 8-item PACES. They will be rated in a 7-point Likert scale (1=positive feelings, 7=negative feelings); but some items will be reverse scored (1=negative feeling, 7=positive feelings). After reverse-scoring the negatively worded items, a higher score will reflect greater enjoyment of physical activity.
Mindful self-care - Psychological health outcome | Collected pre-test, post-test after 16 week intervention program, at 3 months after intervention and at 6 months after intervention.
  Mindful Self-Care Scale - Chinese Version (24 item) measures an individual's level of mindful self-care across various dimensions, including physical care, supportive relationships, mindful awareness, self-compassion and purpose, mindful relaxation, and supportive structure. It is scored in a 5-point Likert scale(0=never, 4=very often). Higher score will indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Ransdell, Professor and Chair, Principal Investigator — Boise State University; Che Hin CHAN, Vice President Chair Professor, Principal Investigator — Education University of Hong Kong; Ng KWOK, Chief Scientist Professor, Principal Investigator — Lithuanian Sports University; Wei Ping TU, Developmental Director, Principal Investigator — ParaVolley Asia Oceania; Paul Lee Hong, Associate Professor, Principal Investigator — University of Southampton; Claudia Wong Ming Yu, Assistant Professor, Principal Investigator — Education University of Hong Kong; Patrick Yung Shu Hang, Professor, Chairman, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- 23 Waterloo Rd, Yau Ma Tei, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Home Affairs Bureau, SAR Government of Hong Kong. A consultancy study on sport for people with disabilities in Hong Kong. Hong Kong: Home Affairs Bureau, SAR Government; 2016.
- [Result] Alvarez K, Salas E, Garofano C. An integrated model of training evaluation and effectiveness. Hum Resour Dev Rev. 2004;3(4):385-416.
- [Result] Lamontagne ME, Arbour-Nicitopoulos KP, Tomasone JR, Cummings I, Latimer-Cheung AE, Routhier F. Translating an evidence-based physical activity service from context to context: a single organizational case study. J Sports Med Ther. 2017;2:39-50.
- [Result] Wong MYC. Translation and validation of the Mindful Self-Care Scale-Chinese Version: a pilot study. Psych. 2020;2(4):338-346.
- [Result] Winnick JP, Short FX. Conceptual framework for the Brockport Physical Fitness Test. Adapt Phys Activ Q. 2005;22(4):323-332.
- [Result] Leung KM, Chu YM, Wong MY. People with Physical Disabilities playing Light Volleyball: A Qualitative Study in Hong Kong. Disability CBR & Inclusive Development. 2020; 31(3):138-150.
- [Result] Leung KM, Chung PK, Chan AWK, Ransdell L, Siu PMF, Sun P, Yang J, Chen TC. Promoting healthy ageing through light volleyball intervention in Hong Kong: study protocol for a randomised controlled trial. BMC Sports Sci Med Rehabil. 2020 Jan 28;12:6. doi: 10.1186/s13102-019-0151-7. eCollection 2020. PMID 32002186
- [Result] Leung KM, Chung PK, Hagger MS. The effects of light volleyball intervention programme in improving selected physical and psychological attributes of older adults in Hong Kong. Int J Sport Exerc Psychol. 2018;18(1):1-12.
- [Result] Zhou Q, Stewart SM, Wan A, Leung CS, Lai AY, Lam TH, Chan SS. Development and Evaluation of a Train-the-Trainer Workshop for Hong Kong Community Social Service Agency Staff. Front Public Health. 2017 Feb 13;5:15. doi: 10.3389/fpubh.2017.00015. eCollection 2017. PMID 28243586
- [Result] Marks B, Sisirak J, Chang YC. Efficacy of the HealthMatters program train-the-trainer model. J Appl Res Intellect Disabil. 2013 Jul;26(4):319-34. doi: 10.1111/jar.12045. Epub 2013 Apr 16. PMID 23589506
- [Result] Damschroder LJ, Reardon CM, Widerquist MAO, Lowery J. The updated Consolidated Framework for Implementation Research based on user feedback. Implement Sci. 2022 Oct 29;17(1):75. doi: 10.1186/s13012-022-01245-0. PMID 36309746
- [Result] Leung KM, Chung PK, Chu W. Evaluation of a sitting light volleyball intervention to adults with physical impairments: qualitative study using social-ecological model. BMC Sports Sci Med Rehabil. 2020 Jul 8;12:41. doi: 10.1186/s13102-020-00187-8. eCollection 2020. PMID 32670590
- [Result] Picorelli AM, Pereira LS, Pereira DS, Felicio D, Sherrington C. Adherence to exercise programs for older people is influenced by program characteristics and personal factors: a systematic review. J Physiother. 2014 Sep;60(3):151-6. doi: 10.1016/j.jphys.2014.06.012. Epub 2014 Aug 3. PMID 25092418
- [Result] Chung PK, Leung KM. Psychometric Properties of Eight-Item Physical Activity Enjoyment Scale in a Chinese Population. J Aging Phys Act. 2018 Oct 12:1-6. doi: 10.1123/japa.2017-0212. Online ahead of print. PMID 29722637
- [Result] Lam CL, Tse EY, Gandek B. Is the standard SF-12 health survey valid and equivalent for a Chinese population? Qual Life Res. 2005 Mar;14(2):539-47. doi: 10.1007/s11136-004-0704-3. PMID 15892443
- [Result] Nettleton B, Smith RG. An approach to the investigation of coincidence anticipation in ball-tracking skills. Percept Mot Skills. 1980 Apr;50(2):676-8. doi: 10.2466/pms.1980.50.2.676. PMID 7375321
- [Result] Katz-Leurer M, Fisher I, Neeb M, Schwartz I, Carmeli E. Reliability and validity of the modified functional reach test at the sub-acute stage post-stroke. Disabil Rehabil. 2009;31(3):243-8. doi: 10.1080/09638280801927830. PMID 18608433
- [Result] Hol AT, Eng JJ, Miller WC, Sproule S, Krassioukov AV. Reliability and validity of the six-minute arm test for the evaluation of cardiovascular fitness in people with spinal cord injury. Arch Phys Med Rehabil. 2007 Apr;88(4):489-95. doi: 10.1016/j.apmr.2006.12.044. PMID 17398251
- [Result] Berg K, Wood-Dauphinee S, Williams JI. The Balance Scale: reliability assessment with elderly residents and patients with an acute stroke. Scand J Rehabil Med. 1995 Mar;27(1):27-36. PMID 7792547
- [Result] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Result] Leung KM, Chung PK, Chu W, Ng K. Physical and psychological health outcomes of a sitting light volleyball intervention program on adults with physical disabilities: a non-randomized controlled pre-post study. BMC Sports Sci Med Rehabil. 2021 Aug 28;13(1):100. doi: 10.1186/s13102-021-00328-7. PMID 34454587
- [Result] Bishop GM, Kavanagh AM, Disney G, Aitken Z. Trends in mental health inequalities for people with disability, Australia 2003 to 2020. Aust N Z J Psychiatry. 2023 Dec;57(12):1570-1579. doi: 10.1177/00048674231193881. Epub 2023 Aug 22. PMID 37606227
- [Result] Buffart LM, Roebroeck ME, Rol M, Stam HJ, van den Berg-Emons RJ; Transition Research Group South-West Netherlands. Triad of physical activity, aerobic fitness and obesity in adolescents and young adults with myelomeningocele. J Rehabil Med. 2008 Jan;40(1):70-5. doi: 10.2340/16501977-0135. PMID 18176740
- [Result] Jung J, Leung W, Schram BM, Yun J. Meta-Analysis of Physical Activity Levels in Youth With and Without Disabilities. Adapt Phys Activ Q. 2018 Oct 1;35(4):381-402. doi: 10.1123/apaq.2017-0123. Epub 2018 Oct 30. PMID 30376716
- See also: Census and Statistics Department, SAR Government of Hong Kong. Persons with disabilities and chronic diseases in Hong Kong. Hong Kong: Census and Statistics Department; Accessed Feb 20, 2022. — https://www.google.com/search?client=firefox-b-d&q=Census+and+Statistics+Department%2C+SAR+Government+of+Hong+Kong.+Persons+with+disabilities+and+chronic+diseases+in+Hong+Kong.+&sei=t-u0aLfwG9u94-EPk8Hs0Q4
- See also: China Disabled Persons' Federation. Statistics on the development of persons with disabilities in 2023. Accessed Feb 20, 2022. — https://english.www.gov.cn/archive/statistics/202405/03/content_WS66349531c6d0868f4e8e6ad9.html
- See also: World Health Organization. WHO guidelines on physical activity and sedentary behaviour: at a glance. Accessed Feb 20, 2022. Published 2020. — https://www.who.int/publications/i/item/9789240015128